CLINICAL TRIAL: NCT03823651
Title: A Research Program Targeting Pre- and Peri-transplant Optimization Program (R-PPOP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00092963
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient (Experimental): These are patients undergoing hematopoetic stem cell transplant. Patients will complete Interval training, undergo psychiatric consult, nutrition/diet evaluation and referral to social worker.
  Interventions: Behavioral: Interval training; Behavioral: Psychiatric consult; Behavioral: Nutrition/diet evaluation; Behavioral: Referral to Social Worker
- Caregiver (Experimental): These are the assigned caregivers for transplant patients. Caregivers will undergo psychiatric consult, nutrition/diet evaluation and referral to social worker.
  Interventions: Behavioral: Psychiatric consult; Behavioral: Nutrition/diet evaluation; Behavioral: Referral to Social Worker

INTERVENTIONS:
Behavioral: Interval training — Patients will be asked to complete up to 3 x 30-minute structured high intensity interval training aerobic exercise sessions/week. For the first session, patients will come to the Duke Center for Living for in person evaluation and training. After the initial training session in person, a subsequent training session will take place at the patient's home via iPad/iPhone videoconference using a device provided to the patient to provide additional support and the opportunity to answer questions. Subsequent sessions will be done independently by patients, but study staff will be available via iPad/iPhone if questions arise.
  Arms: Patient
Behavioral: Psychiatric consult — Subjects who score below threshold on the PHQ2/PHQ9, PC-PTSD/PCL-5, PROMIS-Depression and/or PROMIS-Anxiety assessments will be referred to a psychiatrist for follow up.
Behavioral: Nutrition/diet evaluation — PG-SGA, ASA24, food group tracking Assessments and Vit D, Vit A, albumin, prealbumin, lipids, A1c levels will be used to provide weekly feedback for one month
Behavioral: Referral to Social Worker — Subjects who score below threshold on the PROMIS-Emotional Support and/or PROMIS-Social Isolation assessments will be referred to a social worker for follow up

SUMMARY:
The purpose of this study is to evaluate the feasibility and outcomes of a research pre- and peri-transplant optimization program (R-PPOP) to improve multiple domains of health including physical function, cognitive function, mental health, and diet and nutrition for patients planning to undergo or undergoing hematopoietic stem cell transplantation (HCT).

ELIGIBILITY:
Patient Inclusion Criteria:

* Plan to undergo an allogeneic hematopoietic stem cell transplant for any cancer or non-cancer illness within the next 6 months
* Age 18-80 years

Patient Exclusion Criteria:

* Both patient and caregiver are unable to read and follow directions in English (ok if only patient cannot read and follow directions in English as caregiver will be able to help).
* Any absolute contraindications to exercise:
* recent (< 6 months) acute cardiac event;
* unstable angina;
* uncontrolled dysrhythmias causing symptoms or hemodynamic compromise;
* symptomatic aortic stenosis;
* uncontrolled symptomatic heart failure;
* acute pulmonary embolus;
* acute myocarditis or pericarditis;
* suspected or known dissecting aneurism; or
* coronary artery disease.
* Functional impairment resulting in inability to exercise

Caregiver inclusion criteria

* Identified by patient as their primary caregiver
* Age 18-80 years

Caregiver exclusion criteria

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2024-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Sung, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Adult Bone Marrow Transplant Clinic, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Duke Adult Bone Marrow Transplant program between May 2019 and November 2021. The first subject was consented on May 6, 2019 and the last subject was consented on November 2, 2021.
Pre-assignment Details: 29 subjects (16 patients and 13 caregivers) signed the consent form for this study. 5 subjects (3 patients and 2 caregivers) did not begin the study after signing the consent form. 24 subjects began study activity after signing the consent form.
Period: Overall Study
Arm/Group | Patient | Caregiver
Started | 13 | 11
Completed | 7 | 5
Not Completed | 6 | 6
Not completed — Death | 5 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Caregiver to patient who died | 0 | 5
Not completed — Caregiver to patient who was withdrawn due to physician decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient | Caregiver | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59 (11.6) | 55 (13.8) | 56 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 12
  Male | 10 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 10 | 8 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI (body mass index) [Mean (Standard Deviation); unit: kg/m2] — Population: Caregivers were not included in BMI analysis
  kg/m2
    number analyzed (Participants) | 13 | 0 | 13
    (all) | 29.5 (4.8) |  | 29.5 (4.8)
Weight [Mean (Standard Deviation); unit: kg] — Population: Caregivers not included in weight analysis
  kg
    number analyzed (Participants) | 13 | 0 | 13
    (all) | 90.8 (19.7) |  | 90.8 (19.7)
Diagnosis [Count of Participants; unit: Participants] — Population: Caregivers are not included in the Diagnosis category
  Participants
    number analyzed (Participants) | 13 | 0 | 13
    Myelodysplastic syndrome | 5 |  | 5
    Acute myeloid leukemia | 3 |  | 3
    Diffuse large B-cell lymphoma | 2 |  | 2
    Acute lymphoblastic leukemia | 1 |  | 1
    Chronic lymphocytic leukemia | 1 |  | 1
    Peripheral T-cell lymphoma | 1 |  | 1
Receiving chemotherapy during intervention [Count of Participants; unit: Participants] — Population: Caregivers are not included in the chemotherapy during transplant analysis
  Participants
    number analyzed (Participants) | 13 | 0 | 13
    Yes | 10 |  | 10
    No | 3 |  | 3
Work Status [Count of Participants; unit: Participants]
  Employed Full-Time | 4 | 3 | 7
  Employed Part-Time | 0 | 2 | 2
  Homemaker | 0 | 1 | 1
  Retired | 6 | 4 | 10
  Unemployed/Disabled | 2 | 0 | 2
  Unemployed/Seeking | 0 | 1 | 1
  Unknown/Not Reported | 1 | 0 | 1
Martial Status [Count of Participants; unit: Participants]
  Married or living with significant other | 13 | 10 | 23
  Single, never married | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed at Least Half of Their High Intensity Interval Training Sessions
Description: Participants were asked to record or report their exercise sessions.
Time Frame: 6 months
Population: 13 patients were prescribed the HIIT intervention, but only 9 consistently recorded sessions throughout the duration of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient
Number analyzed (Participants) | 9
Participants | 9

2. Other Pre Specified Outcome: Measuring Changes in the Skin Flora (Microbiome) in Caregivers
Time Frame: baseline, sign off, day 0 (transplant), 7, 14, 21, 30, 60, 90,180, 365
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Changes in Fecal Samples as Measured by 16s rRNA Sequencing in Caregivers
Time Frame: baseline, sign off, day 0 (transplant), 7, 14, 21, 30, 60, 90,180, 365
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Caregiver Quality of Life as Assessed by the Caregiver Strain Questionnaire
Description: Scored as 0 (No, least severe), 1 (Yes, sometimes) and 2 (Yes, on a regular basis, most severe)
Time Frame: 1 year
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Quality of Life as Assessed by the FACT-BMT Questionnaire
Description: Scored from 0 (least severe) to 4 (most severe)
Time Frame: 1 year
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Delirium as Measured by the DOS Assessment
Time Frame: 1 year
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Assessing Falls
Description: Participants will answer Yes/No to whether they have had any falls in the preceding 6 months
Time Frame: 1 year
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Return to Work as Assessed by the Work Assessment
Time Frame: 1 year
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Transplant Length of Stay
Time Frame: 1 year
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Graft Versus Host Disease (GVHD)
Time Frame: 1 year
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Intensive Care Unit Length of Stay
Time Frame: 1 year
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Hospital Length of Stay
Time Frame: 1 year
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Rate of Intensive Care Unit Admission/Re-admission
Time Frame: 1 year
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Rate of Hospital Admission/Re-admission
Time Frame: 1 year
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Rate of Overall Infections
Time Frame: 1 year
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Rate of Fungal Infections
Time Frame: 1 year
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Rate of Viral Infections
Time Frame: 1 year
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Rate of Bacterial Infections
Time Frame: 1 year
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Disease-free Survival
Time Frame: 1 year
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Overall Survival
Time Frame: 1 year
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Changes in Fecal Samples as Measured by 16s rRNA Sequencing in Transplant Patients
Time Frame: baseline, sign off, day 0 (transplant), 7, 14, 21, 30, 60, 90,180, 365, 730
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Measuring Biomarkers of Inflammation/Frailty in Blood Plasma Samples
Description: Biomarker panel to be analyzed: CRP, Eotaxin, Eotaxin-3, FGF (basic), Flt-1/VEGFR-1, GM-CSF, ICAM-1, IFN-γ, IL-10, IL-12/IL-23p40, IL-12p70, IL-13, IL-15, IL-16, IL-17A, IL-17A/F, IL-17B, IL-17C, IL-17D, IL-1RA, IL-1α, IL-1β, IL-2, IL-21, IL-22, IL-23, IL-27, IL-3, IL-31, IL-4, IL-5, IL-6, IL-7, IL-8, IL-8 (HA), IL-9, IP-10, MCP-1, MCP-4, MDC, MIP-1α, MIP-1β, MIP-3α, PlGF, SAA, TARC, Tie-2, TNF-α, TNF-β, TSLP, VCAM-1, VEGF-A, VEGF-C, VEGF-D
Time Frame: 1 year
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Measuring Changes in the Skin Flora (Microbiome) in Transplant Patients
Time Frame: baseline, sign off, day 0 (transplant), 7, 14, 21, 30, 60, 90,180, 365
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Caregiver Support as Assessed by the Caregiver Strain Index Questionnaire
Description: Assessment is scored as 0 (never/least severe), 1 (sometimes), 2 (on a regular basis/most severe)
Time Frame: 1 year
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Social Support as Assessed by the PROMIS Social Isolation Questionnaire
Description: Assessment is scored from 1 (least severe) to 5 (most severe)
Time Frame: 1 year
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Diet as Assessed by the Food Group Tracking Digital Application
Time Frame: 30 days
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Diet as Assessed by the TRU-BMT Digital Application
Time Frame: 30 days
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Nutrition as Assessed by the 24 Hour Food Recall Survey
Time Frame: 30 days
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Mental Health as Assessed by PROMIS Depression Questionnaire
Description: Assessment is scored from 1 (least severe) to 5 (most severe)
Time Frame: 1 year
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Cognitive Function as Assessed by PROMIS Cognitive Questionnaire
Description: Assessment is scored from 5 (least severe) to 1 (most severe)
Time Frame: 1 year
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Physical Function as Assessed by PROMIS Physical Function Questionnaire
Description: Assessment is scored from 5 (least severe) to 1 (most severe)
Time Frame: 1 year
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Physical Activity as Measured by Cardiopulmonary Exercise Testing (CPET)
Description: CPET is scored by measuring changes in V02 max
Time Frame: day 180
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for participants from enrollment through 1 year post-transplant
Description: Adverse events are self-reported by study participants. The patients on this study are undergoing allogeneic stem cell transplantation, which is a procedure that is associated with high rates of adverse outcomes and morbidity. As such, we only record adverse events that are directly reported to us by the study participant or that are directly related to the study activity (i.e. falls during 6 minute walk test, emotional distress from answering study questionnaires, etc.)
Arm/Group | Patient | Caregiver
All-Cause Mortality (participants affected / at risk) | 5/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 2/13 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient (N=13) | Caregiver (N=11)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) — Atrial Fibrillation
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Surgery for hip fracture (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT03823651/Prot_SAP_000.pdf